CLINICAL TRIAL: NCT07130435
Title: The Effect of Nursing Intervention Based on the Salutogenic Model on Sense of Coherence, Healthy Aging, and Quality of Life
Brief Title: The Effect of Salutogenes-Based Nursing Intervention on Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Gülçin Kurt, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-513
Record Dates: First submitted 2025-05-05; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Sense of Coherence
Keywords: Salutogenesis, elderly people, public health nursing
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled intervention using a pretest-posttest experimental design. Participants will be 72 older adults aged 60-70 residing in nursing homes affiliated with the Turkish Ministry of Family and Social Services in Ankara. They will be randomly assigned to either an intervention (n=36) or control (n=36) group. The study aims to evaluate the effect of an intervention based on the salutogenic model on sense of coherence, healthy aging, and quality of life.
Masking Description: No masking will be applied in this study. Both participants and researchers will be aware of the assigned groups due to the nature of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will receive an intervention based on the salutogenic model, aimed at enhancing the sense of coherence and promoting healthy aging. The program will focus on improving participants' overall quality of life by strengthening their internal resources and fostering resilience. The intervention will include educational sessions, guided discussions, and practical strategies for maintaining physical and mental health in older adults with hypertension and diabetes. The intervention will be delivered over a specified period, with regular follow-ups to assess progress.
  Interventions: Behavioral: Salutogenic Model-Based Healthy Aging Program
- control group (No Intervention): Participants in this group will receive standard care as provided by the nursing homes, without any additional intervention based on the salutogenic model. They will continue to receive routine support and healthcare services that are typically available to older adults in the facility, including management of hypertension and diabetes. This group will be monitored for any changes in quality of life and sense of coherence over the course of the study, but no specific program or educational sessions will be provided.

INTERVENTIONS:
Behavioral: Salutogenic Model-Based Healthy Aging Program — The Salutogenic Model-Based Healthy Aging Program is designed to enhance the sense of coherence and promote healthy aging among older adults aged 60-70. The program focuses on strengthening participants' internal resources, building resilience, and improving overall quality of life. It includes educational sessions, group discussions, and practical strategies for managing hypertension and diabetes, all while emphasizing physical, emotional, and mental well-being. The program aims to empower participants to make informed lifestyle choices and cope with the challenges of aging. Participants will receive regular follow-up assessments to track progress and ensure continued support throughout the study period.
  Other Names: educational intervention
  Arms: Intervention Group

SUMMARY:
The world population is rapidly aging, and Turkey is one of the countries where aging is occurring quickly. When the investigators examine the proportion of the elderly population to the total population over the years and decades, the invesitigators observe that the percentage was 3.9% in 1935, 3.4% in 1955, 4.1% in 1975, 5.7% in 2000, 7.2% in 2010, 7.7% in 2013, and 8.5% in 2017. Finally, in 2022, this proportion reached 9.9%. According to population projections, the proportion of the elderly population is expected to be 12.9% in 2030, 16.3% in 2040, 22.6% in 2060, and 25.6% in 2080 (TUIK, 2022).

The ability of elderly individuals to live independently is influenced by their social and economic conditions, physical health, as well as sociodemographic characteristics such as age and gender. The interaction of elderly individuals with society influences their healthy living behaviors. Furthermore, their interaction with personal and societal resources affects their sense of wholeness and quality of life. To achieve a good quality of life, elderly individuals need to use both internal and external resources, and education should support this (Tan et al., 2014). For health services to be effective, they must be sensitive to the differences, experiences, socioeconomic status, and cultural background of individuals. Therefore, health professionals, including nurses, should prioritize providing appropriate health services for elderly individuals during care (Temel et al., 2009). The roles of public health nurses in elderly health include providing education to elderly individuals and caregivers, offering counseling, protecting the health of elderly individuals, conducting physical assessments, teaching self-care and personal hygiene, making home visits when necessary, assessing and taking precautions regarding situations that could cause accidents, evaluating acute health problems and chronic diseases, educating about the management of chronic diseases, and implementing interventions based on nursing diagnoses (Akdemir et al., 2009). The most important principle in ensuring elderly individuals maintain their health and age healthily is to support them in acquiring basic living skills and independence as much as possible. These basic skills, also known as daily living activities, are crucial for preserving the quality of life by enabling elderly individuals to live independently. A review of the literature reveals that there is no evidence of educational or intervention programs aimed at supporting healthy aging for individuals aged 65 and over in Turkey, or programs that focus on holistic health. Therefore, this randomized controlled study will investigate

how an intervention and education program based on the salutogenic model affects elderly individuals' self-efficacy, healthy living behaviors, and coping skills with diseases and stressors. As a result, the applied intervention program will positively impact the quality of life, sense of wholeness, and healthy aging processes of elderly individuals by examining their responses to stressors and revealing the internal and external resources they can utilize.

DETAILED DESCRIPTION:
The world population is rapidly aging, and Turkey is one of the countries where aging is occurring quickly. When the investigators examine the proportion of the elderly population to the total population over the years and decades, the investigators observe that the percentage was 3.9% in 1935, 3.4% in 1955, 4.1% in 1975, 5.7% in 2000, 7.2% in 2010, 7.7% in 2013, and 8.5% in 2017. Finally, in 2022, this proportion reached 9.9%. According to population projections, the proportion of the elderly population is expected to be 12.9% in 2030, 16.3% in 2040, 22.6% in 2060, and 25.6% in 2080 (TUIK, 2022). The increase in the elderly population brings about various health, economic, social, and environmental challenges. In order to address these issues, societies are not only developing care and treatment methods for the elderly but are also giving importance to prevention methods. The ability to live independently is essential for healthy aging and maintaining a healthy population. To support the elderly in living independently, both preventive and therapeutic methods are used. This is because, alongside long life, the quality of life is also of great importance (Gürer et al., 2019). From the perspective of the National Action Plan on Aging, health problems emerge or existing issues are exacerbated with aging, thereby affecting living standards. In addition to the physical changes seen in this period, health problems related to chronic diseases also negatively impact the quality of life.

The increase in life expectancy at birth has contributed to the global increase in the elderly population (onikinciplan.sbb.gov.tr). The ability of elderly individuals to live independently is influenced by their social and economic conditions, physical health, as well as sociodemographic characteristics such as age and gender. The interaction of elderly individuals with society influences their healthy living behaviors. Furthermore, their interaction with personal and societal resources affects their sense of wholeness and quality of life. To achieve a good quality of life, elderly individuals need to use both internal and external resources, and education should support this (Tan et al., 2014). For health services to be effective, they must be sensitive to the differences, experiences, socioeconomic status, and cultural background of individuals. Therefore, health professionals, including nurses, should prioritize providing appropriate health services for elderly individuals during care (Temel et al., 2009). The roles of public health nurses in elderly health include providing education to elderly individuals and caregivers, offering counseling, protecting the health of elderly individuals, conducting physical assessments, teaching self-care and personal hygiene, making home visits when necessary, assessing and taking precautions regarding situations that could cause accidents, evaluating acute health problems and chronic diseases, educating about the management of chronic diseases, and implementing interventions based on nursing diagnoses (Akdemir et al., 2009). The most important principle in ensuring elderly individuals maintain their health and age healthily is to support them in acquiring basic living skills and independence as much as possible. These basic skills, also known as daily living activities, are crucial for preserving the quality of life by enabling elderly individuals to live independently. A review of the literature reveals that there is no evidence of educational or intervention programs aimed at supporting healthy aging for individuals aged 65 and over in Turkey, or programs that focus on holistic health. Therefore, this randomized controlled study will investigate

- Page 2 of 5 [DRAFT] - how an intervention and education program based on the salutogenic model affects elderly individuals' self-efficacy, healthy living behaviors, and coping skills with diseases and stressors. As a result, the applied intervention program will positively impact the quality of life, sense of wholeness, and healthy aging processes of elderly individuals by examining their responses to stressors and revealing the internal and external resources they can utilize. Research Hypotheses Hypothesis 1. H1: There is a difference in the average quality of life scores between elderly individuals in the intervention and control groups. Hypothesis 2. H1: There is a difference in the average sense of wholeness scores between elderly individuals in the intervention and control groups. Hypothesis 2a. H1: There is a difference in the average comprehensibility subscale scores of the sense of wholeness between elderly individuals in the intervention and control groups. Hypothesis 2b. H1: There is a difference in the average meaningfulness subscale scores of the sense of wholeness between elderly individuals in the intervention and control groups. Hypothesis 2c. H1: There is a difference in th

ELIGIBILITY:
Inclusion Criteria:

* Age between 60 and 70 years.

Residing in nursing homes affiliated with the Turkish Ministry of Family and Social Services in Ankara.

A minimum score of 24 on the Mini-Mental State Examination (MMSE).

Diagnosed with Diabetes Mellitus (DM) or Hypertension (HT) for at least the past 3 years.

Exclusion Criteria:

* Known cognitive impairment or difficulty in perception.

Severe hearing or vision impairment.

Inability to participate in the study due to activity intolerance.

Inability to perform daily living activities independently.

Weight loss greater than 3 kg in the past month.

Presence of incontinence.

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — If you plan to analyze the outcomes based on gender (e.g., assessing whether the intervention has a different impact on men vs. women).
Enrollment: 72 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QoL): | Measured at baseline (pre-intervention) and immediately after the intervention (post-intervention).
  The secondary primary outcome will be changes in the participants' quality of life, assessed through a standardized QoL scale, focusing on physical, mental, and social well-being.

OTHER OUTCOMES:
Sense of Coherence (SOC): | Measured at baseline (pre-intervention) and immediately after the intervention (post-intervention).
  The primary outcome measure will be the improvement in participants' sense of coherence, which reflects their ability to manage stress, maintain health, and cope with life's challenges. SOC will be assessed using a validated questionnaire before and after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülçin KURT, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) for this study.